CLINICAL TRIAL: NCT01741337
Title: Central Sleep Apneas Syndrome and Ventricular Function in Patients With Heart Failure, After Coronary Artery Bypass Graft Surgery or Other Coronary Reperfusion
Brief Title: PAC-IC-SAS Pilot Study - Central Sleep Apneas Syndrome and Ventricular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1225; 2012-A01084-39 (Other: ANSM)
Record Dates: First submitted 2012-11-23; First posted 2012-12-04 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Central Sleep Apneas Syndrome; Heart Failure; Coronary Artery Bypass Graft Surgery or Other Coronary Reperfusion
Keywords: central sleep apneas syndrome; heart failure; all coronary reperfusions; adaptive servo-ventilation treatment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients treated by ventilation (Experimental): Adaptive servo-ventilation post-operative treatment for 6 months
  Interventions: Procedure: Adaptive servo-ventilation post-operative treatment for 6 months
- Patients not treated by ventilation (No Intervention): Patients not treated during 6 months by an adaptive servo-ventilation

INTERVENTIONS:
Procedure: Adaptive servo-ventilation post-operative treatment for 6 months
  Other Names: Adaptive servo-ventilation for sleep-disorderd breathing for 6 months
  Arms: Patients treated by ventilation

SUMMARY:
The aim of this clinical trial is to evaluate the effect of an early treatment of sleep-disordered breathing by adaptive servo-ventilation in heart failure patient following coronary artery bypass graft surgery or other coronary reperfusion.

DETAILED DESCRIPTION:
This clinical trial is a pilot study, on patients with central sleep apneas syndrome and heart failure, undergoing coronary artery bypass graft surgery or other coronary reperfusion, and then randomized for the adaptive servo-ventilation treatment application or not after surgery.

The first objective is to evaluate the effect of an early treatment of sleep-disordered breathing by adaptive servo-ventilation in heart failure patient, in terms of ventricular recovery (ejection fraction improvement). This treatment will be instaurated just after coronary artery bypass graft surgery or other coronary reperfusion.

Secondary objectives :

* Assessment of adaptive servo-ventilation effect on the endothelial function, the systemic inflammation and oxidative stress, the insulin resistance, after the surgery in comparison with non treated patient with heart failure and central sleep apneas.
* Assessment of the impact of nocturnal desaturation level on the vascular reactivity and atherosclerosis of mammary vessels collected only during coronary artery bypass graft surgery.
* Assessment of the impact of nocturnal desaturation level on the oxidative stress, inflammation and insulin sensitivity on abdominal and epicardiac adipose tissue collected during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass graft surgery or other coronary reperfusion
* heart failure patient: with altered left ventricular ejection fraction by ultrasonography (45%< LVEF ≤ 50% in 2D) or in 3D
* Patient with central sleep apneas syndrome (SAS)

Exclusion Criteria:

* Aortic or mitral valvular surgery
* Patient already treated for a central SAS
* Patient with an obstructive SAS
* Patient with malignant evolutive pathology
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01-29 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percent of ventricular function recovery (left ventricular ejection fraction) improvement conferred by an adaptive servo-ventilation post-operative treatment | after 6 months of adaptive servo-ventilation post-operative treatment
  Measurement of the left ventricular ejection fraction by a cardiac ultrasonography

SECONDARY OUTCOMES:
Assessment of adaptive servo-ventilation effect on the endothelial function, after the surgery in comparison with non treated patient with heart failure and central sleep apneas. | After 6 months of adaptive servo-sentilation post-operative treatment
  Measurement of peripheral arterial tone
Assessment of the impact of nocturnal desaturation level on the vascular atherosclerosis of mammary vessels collected during coronary artery bypass surgery. | sleep disordered breathing level, 2 months before surgery
  By immunological and histological analysis of mammary vessels
Assessment of the impact of nocturnal desaturation level on the oxidative stress, inflammation and insulin sensitivity of the abdominal and epicardiac adipose tissue collected during surgery. | sleep disordered breathing level, 2 months before surgery
  Measuring inflammatory and oxidative adipose markers
Assessment of adaptive servo-ventilation effect on the systemic inflammation and oxidative stress, the insulin resistance, after the surgery in comparison with non treated patient with heart failure and central sleep apneas. | After 6 months of adaptive servo-sentilation post-operative treatment
  Measurement of inflammatory and oxidative serum markers
Assessment of the impact of nocturnal desaturation level on the vascular reactivity of mammary vessels collected during surgery. | sleep disordered breathing level, 2 months before surgery
  By vascular reactivity study of mammary vessels
Assessment of the impact of nocturnal desaturation level on the abdominal and epicardiac adipose tissue structure collected during surgery. | sleep disordered breathing level, 2 months before surgery
  By immunological and histological analysis of abdominal and epicardiac adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Renaud TAMISIER, MD, PhD, Principal Investigator — University Hospital of Grenoble, France
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Result] Vazir A, Hastings PC, Dayer M, McIntyre HF, Henein MY, Poole-Wilson PA, Cowie MR, Morrell MJ, Simonds AK. A high prevalence of sleep disordered breathing in men with mild symptomatic chronic heart failure due to left ventricular systolic dysfunction. Eur J Heart Fail. 2007 Mar;9(3):243-50. doi: 10.1016/j.ejheart.2006.08.001. Epub 2006 Oct 6. PMID 17030014